CLINICAL TRIAL: NCT02642926
Title: Randomized Controlled Trial Comparing the Efficiency of the Bipolar Energy Compared With the Monopolar Energy in Endometrial Ablation in Women Having Menorrhagia
Brief Title: Comparison of the Efficiency of Bipolar Energy Versus Monopolar Energy in Endometrial Ablation in Women Having Menorrhagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Nazac, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUB-Monobimen
Record Dates: First submitted 2015-12-11; First posted 2015-12-30 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Menorrhagia
Keywords: menorrhagia; higham PBAC score; endometrial ablation; bipolar energy; monopolar energy
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monopolar endoscopic endometrial ablation (Active Comparator)
  Interventions: Procedure: Monopolar current
- Bipolar endoscopic endometrial ablation (Experimental)
  Interventions: Procedure: Bipolar current

INTERVENTIONS:
Procedure: Monopolar current — Hysteroscopic surgical treatment of menorrhagia by use of monopolar current
  Arms: Monopolar endoscopic endometrial ablation
Procedure: Bipolar current — Hysteroscopic surgical treatment of menorrhagia by use of bipolar current
  Arms: Bipolar endoscopic endometrial ablation

SUMMARY:
Since the development a few years ago of bipolar energy in the surgery by operative hysteroscopy, the hysteroscopic treatment of menorrhagia by endometrial ablation can be achieved either by the use of monopolar or bipolar current, in parallel with other techniques labelled as 'second generation' (microwave, radio frequency, thermal destruction ...) treating the uterine cavity.

It seems that the use of the bipolar energy decreases the rate of adhesions but prospective data on the success rate after bipolar endometrial ablation are poor and there is currently no recommendation as to the choice of technique to use. No prospective assessment exists to date in the literature to compare the difference in efficacy on bleedings when using monopolar or bipolar current. The goal of this study is to compare these two energies, by measuring the amount of bleeding calculated by the Higham score 12 months after the intervention.

DETAILED DESCRIPTION:
Menorrhagia are one of the main symptoms that are managed in Gynecology. The evaluation of the volume of menorrhagia is performed by a PBAC score (pictorial bleeding assesment chart). The one described by Higham allows to quantify and qualify periods as being hemorrhagic when the score is above 150.The surgical treatment of choice has long been hysterectomy.

Many studies evaluating the efficacy, safety and cost of different techniques were performed. A recent review of the literature identified eight randomized clinical trials that showed a slight advantage to the hysterectomy, in comparison with the ablation of the endometrium, for the improvement of symptoms and the patient's satisfaction. Hysterectomy is however associated with a longer surgery duration and a longer recovery period. Moreover, most adverse events (major and minor), were significantly more common after hysterectomy.

A retrospective study examined the long-term results of hysteroscopic endometrectomies. During the monitoring, carried out over 4 to 10 years, menorrhagia stopped in 83.4% of cases. Over the same period, 16.6% of the patients had to undergo hysterectomy because menorrhagia had returned.

In terms of cost, one study showed that the total direct and indirect cost of an hysteroscopic treatment of menorrhagia was significantly lower than that of hysterectomies.Endometrial ablation thus offers an alternative to hysterectomy as surgical treatment of menorrhagia.

Several instances and authors recommend this surgery as first line when medical treatment has failed.Initially, the hysteroscopic surgical treatment of menorrhagia was performed by monopolar endoscopic ablation, which requires the use of glycine as a distension medium. Complications proper to the monopolar ablation were described. Because of these complications, the use of bipolar energy has been developped since several years.

Other techniques known 2nd generation techniques have emerged: use of microwave, radio frequency, thermal destruction of the endometrium. They are all comparable in efficiency with a success rate of around 70% with the disadvantage of not having a comprehensive histology and be much more expensive. This diminishes their use because of the cost of purchase of the device.

Although hysteroscopic bipolar ablation is now a routine technique, there are until now no studies in the literature comparing the efficacy of treatment when using monopolar or bipolar energy, for the endometrial resection by hysteroscopy, for menorrhagia management.The goal of this study is to compare these two energies, by measuring the amount of bleeding calculated by the Higham score 12 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from menorrhagia
* Higham score > 150
* No further pregnancy wish
* Failure of a former medical treatment
* Patients consulting a surgeon, for a standard of care surgical intervention

Exclusion Criteria:

* Pregnant women
* Menopausal women
* Patient under anticoagulant treatment, type anti-vitamin K (AVK)
* Patient with a malign endometrial pathology
* Patient with one or several known endo-uterine synechia
* Uterine malformation
* Active and uncured infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Bleeding abundance | 12 months after surgical intervention
  Bleeding abundance will be measured by the Higham score, on a questionnaire sent to the patient.

SECONDARY OUTCOMES:
Bleeding abundance | 6 months after surgical intervention
  Bleeding abundance will be measured by the Higham score, on a questionnaire sent to the patient.
Surgery duration | From the entry till the removal of the hysteroscope from the body -ambulatory surgery (max one day)
  Surgery duration time, measured in minutes. The surgery will be performed according to the standard of care of the hospital, in ambulatory mode.
Per-operative complications rate | From the entry till the removal of the hysteroscope from the body - ambulatory surgery (max one day)
  Number of complications that occured during the surgery duration. The surgery will be performed according to the standard of care of the hospital, in ambulatory mode.
Post-operative complications rate | 6 weeks after the surgical intervention
  Number of complications that occured after the surgery
Re-do surgery rate | 12 months after the surgical intervention
  Re-do surgery rate, because of hysteroscopic treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: André Nazac, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Bicêtre, Kremlin Bicêtre (A.P.H.P), Bicêtre, France

REFERENCES:
- [Background] Duckitt K. Menorrhagia. BMJ Clin Evid. 2015 Sep 18;2015:0805. PMID 26382038
- [Background] Higham JM, O'Brien PM, Shaw RW. Assessment of menstrual blood loss using a pictorial chart. Br J Obstet Gynaecol. 1990 Aug;97(8):734-9. doi: 10.1111/j.1471-0528.1990.tb16249.x. PMID 2400752
- [Background] Fergusson RJ, Lethaby A, Shepperd S, Farquhar C. Endometrial resection and ablation versus hysterectomy for heavy menstrual bleeding. Cochrane Database Syst Rev. 2013 Nov 29;(11):CD000329. doi: 10.1002/14651858.CD000329.pub2. PMID 24288154
- [Background] Boe Engelsen I, Woie K, Hordnes K. Transcervical endometrial resection: long-term results of 390 procedures. Acta Obstet Gynecol Scand. 2006;85(1):82-7. doi: 10.1080/00016340500424314. PMID 16521686
- [Background] Brumsted JR, Blackman JA, Badger GJ, Riddick DH. Hysteroscopy versus hysterectomy for the treatment of abnormal uterine bleeding: a comparison of cost. Fertil Steril. 1996 Feb;65(2):310-6. doi: 10.1016/s0015-0282(16)58091-1. PMID 8566254
- [Background] Mayor S. NICE says hysterectomy must be last option for heavy menstrual bleeding. BMJ. 2007 Jan 27;334(7586):175. doi: 10.1136/bmj.39105.376412.DB. No abstract available. PMID 17255588
- [Background] Berg A, Sandvik L, Langebrekke A, Istre O. A randomized trial comparing monopolar electrodes using glycine 1.5% with two different types of bipolar electrodes (TCRis, Versapoint) using saline, in hysteroscopic surgery. Fertil Steril. 2009 Apr;91(4):1273-8. doi: 10.1016/j.fertnstert.2008.01.083. Epub 2008 Apr 18. PMID 18371962